CLINICAL TRIAL: NCT07234292
Title: Evaluation of Patient Satisfaction With a New Preservative-free Eyelid Cream as a Complementary Care in Post-eyelid Surgery: The ADMIRE Study
Brief Title: Evaluation of Patient Satisfaction With Blephaderm as a Complementary Care in Post-eyelid Surgery.
Status: Not yet recruiting | Type: Observational
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Other Study IDs: LT10100-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Eyelid; Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group receiving Blephaderm
  Interventions: Other: Cosmetic: Blephaderm

INTERVENTIONS:
Other: Cosmetic: Blephaderm — Preservative free eyelid cream: Aqua (water), oleyl erucate, trehalose, sodium acrylates copolymer, lecithin, Ophiopogon japonicus root extract, hydrolyzed hyaluronic acid, maltodextrin, tocopherol, sodium hydroxide, phytic acid, Glycine soja (soybean) oil, Helianthus annuus seed oil.

SUMMARY:
The goal of this non-interventional, open and monocentric study is to evaluate the satisfaction of 30 patients, after 3 months with Blephaderm eyelid cream, as a complementary care in post-eyelid surgery (Blepharopasty or ptosis).

The participant will be asked to use Blephaderm twice a day. The patient satisfaction will be evaluated using a VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients planning a blepharoplasty or a ptosis surgery in at least one eye.
* Patient affiliated to a health social security system
* Female of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end.

Exclusion Criteria:

In terms of population:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Patient who had been deprived of their freedom by administrative or legal decision
* Minor patient.
* Major patient who is under guardianship or who is not able to express his non opposition.
* Patient suspected to be non-compliant according to the investigator's judgment.
* Patient enrolled in another clinical trial or which exclusion period is not over.

In terms of associated pathology

* Patient with a history or active systemic condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk.
* Patient suffering from a severe or progressive disease.
* Patient with known or suspected hypersensitivity to one of the components of the product.

Related to previous or ongoing treatment

* Patient undergoing a topical treatment on the test area or a systemic treatment.
* Patient under a long-term corticosteroid, NSAID or HIV therapy at the investigator appreciation.
* Patient under immunosuppressive therapy
* Patient under bisphosphonate therapy
* Patient having Type 1 diabetes
* Patient having atopic or eczema skin

In terms of lifestyle

* Intensive exposure to sunlight or UV-rays foreseen during the study.
* Patient planning to change her/his life habits during the study.
* Patient with an excessive consumption of alcohol and/or tobacco defined as:
* an excessive consumption of alcohol: Drinking more than
* 4 units a day for adult men and more than 2 units a day for adult women,
* an excessive consumption of tobacco: ≥15-20 Cigarettes Per Day (CPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients undergoing blepharoplasty or ptosis surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
global satisfaction of the patient on eyelid comfort after 3 months of Bllephaderm® use, assessed at M4, using a VAS from 0 (unsatisfied) to 10 (very satisfied). | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre-Vincent Jacomet Private Practice, Paris, France